CLINICAL TRIAL: NCT05627687
Title: Caring Relationships Expression Study (CARES)
Brief Title: Caring Relationships Expression Study
Acronym: CARES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Linda Larkey, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00014913
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Caregiver Burden; Anxiety; Stress
Keywords: Heart Rate Variability; Biofeedback; Alzheimer's disease; Dementia
MeSH Terms: conditions — Caregiver Burden; Anxiety Disorders; Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel randomized controlled trial comparing heart rate variability biofeedback to a music listening control condition, both practiced 4-5 days per week for 8 weeks.
Who Masked: Participant
Masking Description: The participant is advised that they are entering a study in which they will be randomized to one of two conditions designed to potentially reduce stress and caregiver burden. Neither condition is presented as the control, thus participants are blinded to the expectations of the assigned condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening Control (Placebo Comparator): Music listening control (MLC) will consist of listening to selected music tracks of choice using either the Pandora or Spotify app (with coaching to download app and play, and log listening time in diary), specifically choosing a neutral channel, Coffeehouse Playlist. For both interventions, FCG will be asked to practice/listen 10-minutes at a time with their AD patient (sharing as much or as little as is possible/preferred) for at least 4-5 days/week, and asked to complete diary/checklists to show times practicing/listening.
  Interventions: Behavioral: Music Listening Control
- Heart Rate Variability Biofeedback (Active Comparator): Participants will receive coaching in a practice that is guided using an Inner Balance app with a device that senses pulse and provides feedback to help achieve a rhythm of heart rate variability called resonant frequency, or "coherence". They will be guided first in slowed heart-focused breathing and positively-focused emotions and then will connect to the app to receives visual feedback to achieve a favorable HRV.
  Interventions: Behavioral: Heart Rate Variability Biofeedback

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback — Practice using the Inner Balance app and device, 10 minutes/day, 4-5 days per week
  Other Names: Heart Focused breathing
  Arms: Heart Rate Variability Biofeedback
Behavioral: Music Listening Control — Listening to music using the Coffeehouse playlist on either Pandora or Spotify app, 10 minutes/day, 4-5 days per week
  Arms: Music Listening Control

SUMMARY:
This study will examine a heart rate variability biofeedback (HRVB) intervention versus a music listening control (MLC) for 30 family caregivers (FCGs) of Alzheimer's disease (AD) (and related dementias: ADRD) patients to examine feasibility (acceptability/adherence, satisfaction) and direction of change in caregiver burden, stress, resilience, anxiety, self-compassion, and relationship quality over the course of 8-weeks.

DETAILED DESCRIPTION:
This pilot study aims to examine feasibility of implementing a HRVB intervention and an MLC control with AD FCGs. The HRVB and MLC interventions will be evaluated for acceptability (operationalized as adherence to intervention) and satisfaction and to identify necessary intervention modifications. Feasibility benchmarks: 85% of participants will be at least 70% adherent to implementation goals (10-min use 5-7 days per week). Feasibility of randomization will be examined by comparing adherence/retention (expecting similar patterns across interventions). Acceptability/satisfaction with HRVB and MLC will be evaluated in semi-structured interviews post-intervention including detailed probing on feature preferences, barriers/facilitators, suggested improvements for retention.

The second aim of this study is to examine patterns of association of HRVB and MLC with outcomes. The investigators will examine pre- to post-intervention changes (and sustained outcomes at follow-up) in self-reported caregiver burden, stress and resilience. Change in relationship quality will additionally be assessed from pre- to post intervention. Change in ANS balance, a neurophysiological indicator of reduced emotional distress and improved resilience, will be assessed using HRV data at all four timepoints to examine trends and change over time. Significance tests will not be conducted, in alignment with goals for pilot feasibility studies. The investigators will observe the direction of change and outcomes to examine the value of MLC as an appropriate control condition showing minimal placebo effects compared to HRVB.

ELIGIBILITY:
Inclusion Criteria:

* In primary/unpaid FCG role > 6 months
* Caring for mild-to-severe ADRD patient

  * 4 caregiver burden score Own/operate smartphone w data plan

Exclusion Criteria:

* Pacemakers or implanted cardioconverter defibrillator (ICD), or conditions/meds that interfere with HRV measurement/feedback

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale-10 (PSS-10) | Change from baseline to 8 weeks at end of intervention
  10 items describing stress, response format 0-4, total score range 0-40, higher scores indicating worse stress
Caregiver Burden | Change from baseline to 8 weeks at end of intervention
  The Zarit Burden Interview includes 12 items, scoring from 0 to 4 (total range 0 to 48) with higher scores indicating higher perceived caregiver Burden

SECONDARY OUTCOMES:
The Brief Resilience Scale | Change from baseline to 8 weeks at end of intervention
  The Brief Resilience Scale includes 4 items scoring 1-5, total score range, 4-20 with higher scores indicating higher resilience
Self-Compassion Scale | Change from baseline to 8 weeks at end of intervention
  Self-Compassion Scale contains 12 items scoring 1-5, total score range, 12-60 with higher scores indicating higher self-compassion
Relationship Quality | Change from baseline to 8 weeks at end of intervention
  Relationship Quality for caregivers and their caregivee is assessed using 4 items scoring 1-4, total range, 5-20 with higher scores indicating better quality
Depression | Change from baseline to 8 weeks at end of intervention
  Patient Health Questionnaire-4 (PHQ4) using 4 items scoring 0-3, total range 0-12 with higher scores indicating poor mood

CONTACTS AND LOCATIONS:
Overall Officials: Linda K Larkey, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University Downtown Campus, Phoenix, Arizona, United States